CLINICAL TRIAL: NCT00491218
Title: The Addition of Cardiac Computed Tomography to Exercise Treadmill Testing in the Evaluation of Angina
Brief Title: The Addition of Cardiac CT to Exercise Treadmill Testing in the Evaluation of Angina
Acronym: CT-EXTRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Other Study IDs: 07-12030
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Angina
Keywords: impact of cardiac computed tomography on outpatient angina evaluation; downstream resource utilization
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The current outpatient evaluation for angina in low and intermediate risk patients typically starts with a functional assessment for coronary ischemia. Exercise treadmill testing is often selected as the initial diagnostic modality for coronary artery function. However, exercise treadmill testing is limited by its moderate sensitivity and specificity, often resulting in further cardiac resource utilization for patient risk stratification and reassurance. With the advent of coronary multislice computed tomography (MSCT) angiography, coronary artery anatomy can now be evaluated noninvasively. Despite its impressive performance characteristics, the role of coronary MSCT angiography in the outpatient evaluation of angina remains undefined.

CT-EXTRA compares the impact on patient safety and downstream resource utilization of a novel initial diagnostic strategy employing the addition of coronary MSCT angiography to exercise treadmill testing with a standard diagnostic strategy of exercise treadmill testing for the ambulatory evaluation of low-intermediate risk patients with possible angina. The study is a single center, prospective, non-blinded, randomized clinical trial. Men and women, age 18-70, with a low to intermediate pretest probability of coronary artery disease who are referred for an exercise treadmill test for angina are eligible. Subjects are randomized either to an initial diagnostic strategy of exercise treadmill testing or exercise treadmill testing with coronary MSCT angiography. Subsequent diagnostic testing and treatment are the discretion of the referring physician. Subjects will be clinically followed for 24 months.

The clinical impact on patient safety and downstream clinical resource utilization of this novel diagnostic strategy in which both coronary artery anatomy and function are initially evaluated will be determined. The primary outcome is a composite endpoint consisting of freedom from adverse cardiac events, further cardiac diagnostic testing, and future cardiac clinical encounters. Secondary outcomes include the impact on the indiscriminate use of coronary angiography, subject anxiety, depression, motivation for healthy behavioral change, and satisfaction with diagnostic evaluation and use of antiplatelet and antilipid therapy. Lastly, the cost effectiveness of the routine addition of coronary MSCT angiography in the outpatient evaluation of possible angina will be determined.

DETAILED DESCRIPTION:
CT-EXTRA is a randomized clinical trial that will compare a novel diagnostic strategy employing the addition of coronary MSCT angiography to exercise treadmill testing with a standard diagnostic strategy of exercise treadmill testing for the outpatient evaluation of low-intermediate risk patients with possible angina. This is the first randomized clinical trial that evaluates a diagnostic strategy for outpatient chest pain that incorporates a noninvasive assessment of both coronary artery function and anatomy. CT- EXTRA will determine whether coronary MSCT angiography adds any incremental prognostic value over exercise treadmill testing alone for predicting future adverse cardiac events and reduces downstream clinical resource utilization. This study will also evaluate the impact of this strategy on the avoidance of unnecessary invasive coronary angiography, statin and aspirin prescription, patient anxiety, satisfaction with the diagnostic approach, and motivation for healthy behavioral change. Finally, an economic analysis will be performed to assess the differences in overall healthcare costs between the diagnostic approaches. In today's managed care-dominated paradigm, it is paramount that a new diagnostic modality such as coronary MSCT angiography is not only clinically effective but cost effective as well. CT EXTRA will provide critical information to clinicians and health care administrators on the clinical and cost effectiveness of an initial diagnostic strategy employing routine coronary MSCT angiography in the evaluation of patients for possible angina.

300 male and female military health care beneficiaries between the ages of 18-70, who are low to intermediate risk for symptomatic coronary artery disease and are referred to the Walter Reed Cardiology Clinic for an exercise treadmill test for the evaluation of possible angina (chest pain or angina-equivalent).

This study is a randomized, non-blinded, prospective trial to be conducted in the Cardiology clinic at Walter Reed Army Medical Center. Patients, age 18-70 years, referred to the Cardiology clinic for an exercise treadmill test for an outpatient evaluation of possible angina and are low-intermediate risk for symptomatic coronary artery disease, will be eligible. All patients who meet the aforementioned inclusion/exclusion criteria will be consented by an investigator and randomized from sealed envelopes to either "mandatory coronary MSCT angiography" or "no coronary MSCT angiography" before initiation of exercise treadmill testing. The randomization sequence will be generated using a sequence of computer-generated random numbers. All consented subjects will complete surveys assessing baseline depression using the Beck Depression Inventory, anxiety using the State and Trait Anxiety Inventory, and motivation healthy behavioral change using the ladder scale questionnaire. Completion of these three questionnaires are for research purposes and will take approximately 15 minutes.

Exercise Treadmill Testing

All subjects will undergo exercise treadmill testing as initially ordered by the referring physician. All exercise treadmill testing will be conducted at the Cardiology clinic at Walter Reed Army Medical Center according to standard clinic protocol. Testing will be conducted by a health care professional (staff physician, fellow, or nurse practitioner) not associated with the protocol. A Cardiology staff physician not affiliated with the protocol will officially interpret each exercise treadmill test. Subjects will perform a graded exercise treadmill test according to a Full Bruce protocol aimed at reaching 85% of the maximal predicted heart rate for age. According to standard clinical practice, an exercise treadmill test is considered positive if 0.1 mV of new horizontal or downsloping ST segment depression or ST segment elevation 0.80 ms beyond the J point occurs during exercise or recovery in two or more contiguous lead. A nondiagnostic test is defined as the absence of ischemic electrical changes in the setting of reproduction of chest pain symptoms or when peak heart rate is ≤85 % of the age-predicted maximal heart rate. An exercise treadmill test is considered negative when > 85% of the age-predicted maximal heart rate is achieved and reproduction of anginal symptoms and development of electrocardiographic ischemic changes are absent. In accordance with standard clinical practice, exercise treadmill testing will be prematurely terminated in the event of lightheadedness, severe ST depression (>2mm) or elevation (>1mm), ventricular or supraventricular arrhythmias, exaggerated blood pressure increase (>250 mm Hg systolic or >120mm Hg diastolic) and a >10mm Hg decrease in diastolic blood pressure. Upon completion of exercise treadmill testing, the subject will be provided a copy of the results and official interpretation of the exercise treadmill test for inclusion in their medical records. A copy of the exercise treadmill test results will be kept in the subject's file for the investigational team. Completion of an exercise treadmill test generally takes about 25 minutes.

Immediately Following Exercise Treadmill Testing

All consented subjects following exercise treadmill testing will undergo initial laboratory assessment to include fasting lipid panel (LDL-C, HDL-C, and triglycerides), C-reactive protein, fasting blood glucose, creatinine, thyroid stimulating hormone (TSH) and urine pregnancy test (for females). Approximately 15 mL (3 teaspoons) of blood will be drawn by the central laboratory, the clinical laboratory at Walter Reed Army Medical Center. Excess blood will be discarded by the central laboratory according to their standard protocol. All laboratory values will be processed through this central laboratory.

Subjects assigned to the "no coronary MSCT angiography" arm will follow up with their referring physician for further evaluation. Additional selection of testing, consultation, and choice of therapy is at the discretion of the referring physician. Coronary CT angiography will not be available to this group of subjects. Otherwise, the protocol will not predetermine the clinical diagnostic or treatment course for the subject. This approach will simulate the previous standard of care for the evaluation of possible angina (prior to the availability of coronary CT angiography in clinical practice). By excluding the option of coronary CT angiography in this group, any possible incremental value of the test can more accurately be assessed.

In the event of a "high risk" exercise treadmill test, subjects will be offered inpatient admission. High risk tests will include any of the following: the occurrence of sustained ventricular tachycardia, syncope, a high risk Duke treadmill score (>-10), limiting angina in stage 1 of the Full Bruce protocol, > 2 mm ST depression in 3 or more leads in stage 1 of the Full Bruce protocol. Subjects with such high risk tests who are assigned to the "no coronary MSCT angiography" arm will be encouraged to undergo invasive coronary angiography. Subjects assigned to the "mandatory coronary MSCT angiography" arm will undergo coronary MSCT angiography in an expedited manner. This will be followed by invasive coronary angiography, if warranted, 48 hours later. Because the protocol excludes subjects deemed as having a high pretest probability of obstructive coronary artery disease, the potential for this occurrence should be minimized.

Patients assigned to the "mandatory coronary MSCT angiography" arm will be scheduled for coronary MSCT angiography on an outpatient basis. The procedure for coronary MSCT angiography is described below. After completion of coronary MSCT angiography, the results will be provided to the referring physician. Additional selection of testing, consultation, or therapy is at the discretion of the referring physician. The protocol will not predetermine the clinical course for the subject following coronary MSCT angiography.

Coronary MSCT angiography

Pre-procedural Medications: In order to obtain high quality computed tomographic images with minimal motion artifacts, the goal heart rate is ≤ 65 beats per minute. This usually requires administration of beta-blocker medications before image acquisition. In addition, subjects with baseline low rates (> 65bpm) generally need a reduced dose of beta-blockers to blunt increases in rate during the MSCT scan due to anxiety and or reflex responses to contrast. The dose of initial oral beta-blocker will be determined based on resting heart rate at the time of exercise treadmill testing. For subjects with a baseline heart rate above 65bpm and blood pressure above 100/50, 100-150mg of short acting metoprolol will be prescribed by the investigator. Subjects will be instructed to ingest this medication approximately one hour before the scheduled outpatient MSCT scan. For subjects with heart rates above 50bpm and less than 65bpm and blood pressure above 100/50, 25-50 mg of oral short acting metoprolol will be prescribed by the investigator. Subjects will be instructed to ingest this medication approximately one hour before the scheduled outpatient MSCT scan. For subjects with a baseline heart rate < 50bpm, no metoprolol will be prescribed.

On the day of the MSCT scan and upon arrival to the Radiology Department, the subject will receive a peripheral upper extremity intravenous catheter, placed by a certified nurse in the Radiology Department. The subject's baseline blood pressure and heart rate will be recorded. For subjects whose heart rate remains ≥ 65 beats per minute and blood pressure ≥ 100/50, intravenous metoprolol (5 mg aliquots every 2-5 minutes under close observation and continuous telemetric monitoring, up to 40 mg total) will be administered by a cardiology staff or fellow. Once satisfactory heart rate and blood pressure stability are established, subjects will undergo MSCT testing as listed below. However, if target heart rate is not achievable by this protocol, this is not cause for exclusion from the study, since feasibility and accuracy studies have shown that diagnostic scans can be obtained in many patients with higher heart rates with advanced scanners. Nitroglycerin, a coronary vasodilator, will be administered to all subjects (0.8 mg sublingually) approximately 1 minute before initiation of the MSCT scan to optimize image quality. Subjects will be queried regarding the recent use (within the previous 72 hours) of medications for erectile dysfunction (Cialis, Levitra and Viagra) on the day of the MCST scan since these drugs can interact with nitroglycerin to cause a potential life-threatening hypotensive effect. On the day of the scheduled MSCT scan, subjects who admit to have taken Cialis within the past 72 hours or Levitra / Viagra within the past 48 hours will not be allowed to undergo coronary MSCT angiography and will be rescheduled. Subjects will be instructed to withhold these medications for at least 3 days before the scheduled scan.

All female subjects who are randomized to the MSCT arm will be required to wear a radioprotective bismuth shield during the actual MSCT scan. This radioprotective brassiere (Cone Instruments Inc, Solen, Ohio) composed of neoprene and bismuth trioxide has been studied in 16 slice CT scans and has been shown to reduce breast radiation exposure by approximately 40%.25 The bra will be placed directly over both breasts of the female subjects by either a female nurse or technician in the Radiology Department. The adhesive strips on the undersurface of these radioprotective bras will prevent any slippage during the actual scan. Depending on the bust size of the subject, either a medium or large bra will be employed for best fit. Each bra is intended for single patient use only and will be discarded after each study. The effect of these bismuth shields on image interpretation is unknown. If images of the coronary arteries are deemed to be unevaluable, women 40 years and younger will be excluded from participation in the study. In this event, only women greater than the age of 40 years will be enrolled and radioprotective shields will not be used.

Subject follow-up

After completion of initial testing (exercise treadmill test +/- MSCT angiography), subjects will be returned to the referring physicians who will dictate further clinical management. The results of the exercise treadmill testing and coronary MSCT angiography (if applicable) will be provided to the referring physician. Additional selection of testing, consultation, and choice of therapy is at the discretion of the referring physician. For subjects assigned to the "no coronary MSCT angiography" arm, the referring provider will be instructed not to make MSCT an available option for these subjects if further testing is deemed appropriate. Otherwise, the protocol will not predetermine the clinical diagnostic or treatment course for the subject. This approach should simulate actual clinical practice and the previous standard of care (prior to availability of MSCT) and will allow assessment of downstream clinical resource utilization in an unbiased fashion.

Subjects will be followed for a total of two years. During that time, the following factors will be evaluated:

* Status of the presenting syndrome including final diagnosis
* Number of cardiac visits to an outpatient physician or emergency department (ED) because of chest pain/anginal equivalent
* Cardiac hospitalizations for chest pain syndrome/angina equivalent
* Requirement for additional cardiac diagnostic testing, namely further stress testing (nuclear, MRI, echocardiography) and/or cardiac catheterization
* Need for additional radiographic testing for incidental findings found on coronary MSCT
* Need for coronary revascularization procedures
* Unstable angina, myocardial infarction or cardiac death. Myocardial infarction is defined as a cardiac event requiring admission to the hospital with the development of cardiac enzyme level elevation. Unstable angina is defined by accelerating anginal symptoms with or without ischemic electrocardiographic changes requiring hospital admission and coronary revascularization. Death will be attributed to a cardiac origin in the case of documented significant arrhythmia and/or cardiac arrest, congestive heart failure, or myocardial infarction. Moreover, any unexplained death that occurs suddenly out of the hospital will be ascribed a cardiac cause.
* Prescription of antilipid and antiplatelet therapy

These factors will be determined by electronic medical record review (CHCS-II) and telephonic interview with the subjects every 6 months for a total of 2 years. Any visit to an outpatient clinic or ED and any inpatient admission will be categorized as "cardiac" if the presenting complaint is chest pain or identical to the original complaint which prompted the initial exercise treadmill test referral.

Subjects will return to the clinic at 12 months to complete questionnaires to assess changes in depression, anxiety and motivation for healthy behavioral change using the Beck Depression Inventory(BDI), State and Trait Anxiety Inventory (STAI) and ladder scale respectively. Subjects will also be surveyed about their current perception of chest pain as cardiac or noncardiac and the utility of their index cardiovascular evaluation, to provide insight into the etiology of their symptoms.

Endpoints Primary The primary outcome will be a composite endpoint consisting of adverse cardiac events and cardiac resource utilization. Specifically, this will include the occurrence of adverse cardiac events (cardiac death, myocardial infarction, unstable angina, coronary revascularization), utilization of additional diagnostic testing for initial complaint, and the occurrence of future clinical outpatient/inpatient/ED encounters for the initial cardiac complaint.

Secondary

Secondary endpoints will include:

1. Occurrence of adverse cardiac events (cardiac death, myocardial infarction, unstable angina, coronary revascularization)

. 2. Need for subsequent cardiac diagnostic testing for the initial complaint of angina/angina equivalent 3. Occurrence of future clinical outpatient/inpatient/ED encounters for the initial cardiac complaint 4. Avoidance of unnecessary cardiac catheterizations 5. Change in motivation for healthy behavioral change, as assessed by the ladder motivational scale 6. Change in subject anxiety, as assessed by the State and Trait Anxiety Inventory.

7. Change in subject depression, as assessed by the Beck Depression Inventory. 8. Satisfaction with diagnostic evaluation for initial complaint

Predefined Analyses

In addition to the primary and secondary outcomes, there will be two predefined analyses related to these outcomes.

1. Cost Efficiency Analysis, measured as total direct per-patient cost incurred for each diagnostic strategy as related to the primary outcome. The direct per -patient cost in the evaluation of outpatient angina will be calculated by adding the following components and dividing by the number of patients tested:

1. cost of all initial tests of each diagnostic arm (exercise treadmill testing +/- coronary MSCT angiography
2. cost of any additional cardiac diagnostic tests deemed necessary by the referring provider after the completion of the initial diagnostic strategy arms for evaluation of the initial complaint
3. cost of any subsequent inpatient/outpatient/ED evaluations for the initial cardiac complaint over the following 24 months
4. cost of any subsequent radiographic testing needed for incidental findings found on MSCT over the following 24 months The cost of the different diagnostic tests utilized (coronary MSCT angiography, exercise treadmill testing, myocardial perfusion testing, exercise echocardiography, coronary angiography, and other radiographic tests) and clinical encounters (inpatient admissions, ED evaluations, outpatient evaluations) will be estimated from current Medicare reimbursement rates.

2. Statin and aspirin use, measured as the change in the prevalence of statin and aspirin use among subjects in each diagnostic arm.

ELIGIBILITY:
Inclusion Criteria:

1. Chest pain or anginal equivalent symptoms possibly suggestive of symptomatic coronary artery disease.
2. Low-intermediate risk (<75% pretest probability) for symptomatic coronary artery disease on basis of age, sex, and quality of reported symptom as classified by the Diamond and Forrester scheme6
3. Referred to Walter Reed Cardiology clinic for an exercise treadmill test as the initial diagnostic test of choice
4. Age equal to or greater than 18 years and less than 70 years
5. Ability to provide informed consent

Exclusion Criteria:

1. Abnormal baseline electrographic changes that would preclude proper diagnosis of ischemia including preexcitation (Wolff-Parkinson-White) syndrome, a paced ventricular rhythm, more than 1 mm of ST depression at rest, complete left bundle branch block, or criteria for left ventricular hypertrophy, even if they have less than 1 mm of baseline ST depression
2. Presence of known pre-existing coronary artery disease (known prior myocardial infarction, EKG evidence of prior infarction, prior angiographic evidence of significant coronary artery disease, history of prior coronary revascularization).
3. Previous outpatient or inpatient evaluation for coronary artery disease to include exercise treadmill testing, stress echocardiography or nuclear myocardial perfusion studies within the last three years.
4. Presence of signs or symptoms that are clearly compatible with non-cardiac chest pain, including musculoskeletal, gastrointestinal or neuropathic causes.
5. Renal insufficiency (creatinine >1.5mg/dl) or renal failure requiring dialysis.
6. Baseline heart rate > 100bpm, atrial fibrillation or other markedly irregular rhythm (frequent ectopy, multifocal atrial tachycardia) on baseline ECG.
7. Pregnancy or unknown pregnancy status.
8. Known allergy to iodinated contrast.
9. Inability to tolerate beta-blocking drugs, including patients with reactive airways disease requiring maintenance inhaled bronchodilators or steroids, complete heart block or second-degree atrioventricular block.
10. Patients with hyperthyroidism including Grave's disease and toxic multinodular goiter
11. Computed tomography imaging, or iodinated contrast administration over 50 ml, within the past 48 hours.
12. Unwillingness to withhold ingestion of metformin or commonly used erectile dysfunction medications (Viagra, Cialis, Levitra) for 48 hours prior to MSCT scan.
13. Previous history of radiation therapy to the thorax.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-06

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Devine, MD, Principal Investigator — WRAMC Cardiology
Locations (1):
- Walter Reed Army Medical Center Cardiology Service, Washington D.C., District of Columbia, United States